CLINICAL TRIAL: NCT05556616
Title: A Phase 1b Open-label Study to Evaluate the Safety and Tolerability of Intravenous Modakafusp Alfa as Part of Combination Therapy in Adult Patients With Multiple Myeloma
Brief Title: A Study of Modakafusp Alfa in Adult Participants With Multiple Myeloma
Acronym: iinnovate-2
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Due to strategic reasons (no safety concerns).
Sponsor: Teva Branded Pharmaceutical Products R&D LLC (Industry)
Responsible Party: Sponsor
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TAK-573-1502; 2022-001418-20 (EudraCT Number)
Record Dates: First submitted 2022-09-23; First posted 2022-09-27 (Actual); Results first posted 2025-08-06 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Multiple Myeloma
Keywords: Drug Therapy
MeSH Terms: conditions — Multiple Myeloma | interventions — Lenalidomide; Bortezomib; carfilzomib; daratumumab; pomalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Group 1 (NDMM): Modakafusp Alfa 80 mg + Lenalidomide 10 mg (Experimental): Participants received 80 milligrams (mg) modakafusp alfa, infusion intravenously (IV), once on Day 1, once every 4 weeks (Q4W), in combination with 10 mg lenalidomide capsules orally once daily continuously on Days 1 to 28, in a 28-day (4-week) treatment cycle until disease progression, unacceptable toxicity, or to a maximum of 2 years for measurable/minimal residual disease-negative (MRD [-]) participants, whichever occurred first.
  Interventions: Drug: Modakafusp alfa; Drug: Lenalidomide
- Group 2 (RRMM Doublets): Modakafusp Alfa 80 mg + Pomalidomide 2 mg (Experimental): Participants received 80 mg modakafusp alfa, infusion IV, once on Day 1, Q4W in combination with 2 mg pomalidomide capsules orally once daily on Days 1 to 21 in a 28-day (4-week) treatment cycle until disease progression, unacceptable toxicity, or until any other discontinuation criterion was met, whichever occurred first.
  Interventions: Drug: Modakafusp alfa; Drug: Pomalidomide
- Group 2 (RRMM Doublets): Modakafusp Alfa 80 mg + Pomalidomide 4 mg (Experimental): Participants received 80 mg modakafusp alfa, infusion IV, once on Day 1, Q4W in combination with 4 mg pomalidomide capsules orally once daily on Days 1 to 21 in a 28-day (4-week) treatment cycle until disease progression, unacceptable toxicity, or until any other discontinuation criterion was met, whichever occurred first.
  Interventions: Drug: Modakafusp alfa; Drug: Carfilzomib
- Group 2 (RRMM Doublets): Modakafusp Alfa 80 mg + Carfilzomib 20/70 mg/m^2 (Experimental): Participants received 80 mg modakafusp alfa, infusion IV, once on Day 1, Q4W in combination with 20/70 milligrams per meter square (mg/m^2) carfilzomib IV, on Day 1, 8 and 15 of a 28-day (4-week) treatment cycle until disease progression, unacceptable toxicity, or until any other discontinuation criterion was met, whichever occurred first.
  Interventions: Drug: Modakafusp alfa; Drug: Bortezomib
- Group 2 (RRMM Doublets) Arm 4: Modakafusp alfa + Bortezomib (Experimental): Participants were planned to receive modakafusp alfa, infusion IV, once on Day 1, Q4W in combination with bortezomib injection subcutaneously on Days 8, 15, and 22 for the first 8 cycles and subsequently on Days 8 and 22 of a 28-day (4-week) treatment cycle until disease progression, unacceptable toxicity, or until any other discontinuation criterion is met, whichever occurs first.
  Interventions: Drug: Modakafusp alfa; Drug: Bortezomib; Drug: Pomalidomide
- Group 3 (RRMM Triplets) Arm A: Modakafusp alfa + Pomalidomide + Bortezomib (Experimental): Participants were planned to receive modakafusp alfa, infusion IV, once on Day 1, Q4W in combination with pomalidomide capsules orally once daily on Days 1 to 21 in a 28-day (4-week) treatment cycle along with bortezomib injection subcutaneously on Days 8, 15 and 22 for the first 8 cycles and subsequently on Days 8 and 22 of a 28-day (4-week) treatment cycle until disease progression, unacceptable toxicity, or until any other discontinuation criterion is met, whichever occurs first.
  Interventions: Drug: Modakafusp alfa; Drug: Bortezomib; Drug: Pomalidomide
- Group 3 (RRMM Triplets) Arm D: Modakafusp alfa + Daratumumab + Pomalidomide (Experimental): Participants were planned to receive modakafusp alfa, infusion IV, once on Day 1, Q4W in combination with daratumumab injection subcutaneously on Days 1, 8, 15 and 22 of Cycles 1 and 2, further followed by on Days 1 and 15 of Cycles 3 to 6, thereafter on Day 1 on a 28-day (4-week) treatment cycle along with pomalidomide capsules orally once daily on Days 1 to 21 in a 28-day (4-week) treatment cycle until disease progression, unacceptable toxicity, or until any other discontinuation criterion is met, whichever occurs first.
  Interventions: Drug: Modakafusp alfa; Drug: Daratumumab; Drug: Pomalidomide

INTERVENTIONS:
Drug: Modakafusp alfa — Modakafusp alfa intravenous infusion.
  Other Names: TAK-573
Drug: Lenalidomide — Lenalidomide capsules orally.
  Arms: Group 1 (NDMM): Modakafusp Alfa 80 mg + Lenalidomide 10 mg
Drug: Bortezomib — Bortezomib injection subcutaneously.
  Arms: Group 2 (RRMM Doublets) Arm 4: Modakafusp alfa + Bortezomib; Group 2 (RRMM Doublets): Modakafusp Alfa 80 mg + Carfilzomib 20/70 mg/m^2; Group 3 (RRMM Triplets) Arm A: Modakafusp alfa + Pomalidomide + Bortezomib
Drug: Carfilzomib — Carfilzomib intravenous infusion.
  Arms: Group 2 (RRMM Doublets): Modakafusp Alfa 80 mg + Pomalidomide 4 mg
Drug: Daratumumab — Daratumumab injection subcutaneously.
  Arms: Group 3 (RRMM Triplets) Arm D: Modakafusp alfa + Daratumumab + Pomalidomide
Drug: Pomalidomide — Pomalidomide capsules orally.
  Arms: Group 2 (RRMM Doublets) Arm 4: Modakafusp alfa + Bortezomib; Group 2 (RRMM Doublets): Modakafusp Alfa 80 mg + Pomalidomide 2 mg; Group 3 (RRMM Triplets) Arm A: Modakafusp alfa + Pomalidomide + Bortezomib; Group 3 (RRMM Triplets) Arm D: Modakafusp alfa + Daratumumab + Pomalidomide

SUMMARY:
The main aims of this study are to test for any side effects from modakafusp alfa in combination therapy and to determine the recommended dose of combination therapy with modakafusp alfa. The dose of modakafusp alfa will be increased a little at a time until the highest dose that does not cause harmful side effects is found. Participants will be given modakafusp alfa through a vein.

DETAILED DESCRIPTION:
The drug being tested in this study is called modakafusp alfa (TAK-573). The study will evaluate the safety, tolerability and determine the recommended dose of modakafusp alfa in combination with lenalidomide in participants with multiple myeloma (MM), or in combination with pomalidomide, bortezomib, carfilzomib, or daratumumab in participants with relapsed/refractory multiple myeloma (RRMM).

The study consists of 3 Groups: Group 1: MM Maintenance Therapy, Group 2: RRMM Doublets, Group 3: RRMM Triplets.

The study will enroll approximately 18 participants in Group 1, 66 in Group 2, and 36 in Group 3. Participants will be assigned to one of the following treatment groups as given below:

* Group 1 (MM Maintenance) Arm 1: Modakafusp alfa + Lenalidomide
* Group 2 (RRMM Doublets) Arm 2: Modakafusp alfa + Pomalidomide
* Group 2 (RRMM Doublets) Arm 3: Modakafusp alfa + Bortezomib
* Group 2 (RRMM Doublets) Arm 4: Modakafusp alfa + Carfilzomib
* Group 3 RRMM Triplets) Arm A: Modakafusp alfa + Pomalidomide + Bortezomib
* Group 3 (RRMM Triplets) Arm D: Modakafusp alfa + Daratumumab + Pomalidomide

Group 2 Arm 4 is closed for enrollment.

The study will be conducted worldwide. The maximum treatment duration in this study for Group 1 is until disease progression or unacceptable toxicity, or up to 2 years for minimal/measurable residual disease (MRD) negative [-] participants, whichever occurs first. The maximum treatment duration in this study for Group 2 and Group 3 is until disease progression, unacceptable toxicity or until any other discontinuation criterion is met, whichever occurs first. Overall time to participate in the study is approximately up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

1. Group 1 (MM maintenance: modakafusp alfa/lenalidomide) only must have:

   1. MM based on standard IMWG diagnostic criteria.
   2. Undergone autologous stem cell transplantation (ASCT) for the treatment of MM within 12 months of the start of induction therapy and completed ASCT within 180 days before enrollment- (regardless of the lines of treatment).Consolidation cycles are allowed. Tandem transplant is allowed.
   3. Not started lenalidomide maintenance before enrollment. Time to initiation of maintenance therapy: participants may start maintenance therapy as early as 60 days after transplantation and up to 180 days after transplantation or consolidation.
   4. MRD positive ( after ASCT (MRD assessed at a threshold of 10^-5 by local standard-of-care (SOC) methods or central assessment, if a prior local MRD assessment had not been performed).
   5. No prior progression after initial therapy (at any time before starting maintenance). Participants whose induction therapy was changed due to suboptimal response or toxicity will be eligible if they do not meet criteria for progression. In addition, no more than 2 regimens will be allowed before ASCT, excluding dexamethasone alone.
   6. No prior allogeneic hematopoietic stem cell transplant or solid organ transplant.
   7. Recovered to Grade less than or equal to (<=) 1 ASCT-related toxicities from the reversible effects of ASCT (except for alopecia and amenorrhea). MM based on standard IMWG diagnostic criteria.
2. Groups 2 and 3 (RRMM doublets and RRMM triplets) must have:

   1. Measurable disease, defined as at least 1 of the following:

      * Serum M-protein >=0.5 g/dL (>=5 g/L) on serum protein electrophoresis (SPEP).
      * Urine M-protein >=200 mg/24 hours on urine protein electrophoresis (UPEP).
      * Serum free light chain (FLC) assay result with an involved FLC level >=10 mg/dL (>=100 mg/L), provided the serum FLC ratio is abnormal (per IMWG criteria).
   2. A confirmed diagnosis of MM according to International Myeloma Working Group (IMWG) criteria with documented disease progression in need of additional therapy as determined by the investigator.
   3. For Group 2 RRMM doublet arms only: Participants who have received at least 3 prior lines of antimyeloma therapy, including at least 1 proteosome inhibitor (PI), 1 immunomodulatory drug (IMiD) and 1 anti-CD38 monoclonal antibody (mAb) drug, or who are triple refractory to a PI, and IMiD, and an anti-CD38 mAb drug regardless of the number of prior line(s) of therapy.

   d. For Group 3 RRMM triplet arms only: Participants who have received 1 to 3 prior lines of antimyeloma therapy including at least 1 PI and, 1 IMiD, and who are not refractory to the combination partners.

   e) For anti-CD38 arms, forced expiratory volume in 1second (FEV1) >=50% predicted by pulmonary function testing.
3. Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2 at screening
4. Has adequate organ function at screening as determined by the laboratory values required for enrollment: Absolute neutrophil count (ANC) >=1000 per cubic millimeter (/mm^3) (or >=1*10^9/L); Platelets >=75,000/mm^3 (>=75*10^9/L); Hemoglobin >=8.0 g/dL; estimated creatinine clearance >=30 mL/min (Cockcroft-Gault formula); Total serum bilirubin <=2.0*Upper limit of normal (ULN); an exception for participants with Gilbert's syndrome may be granted after discussion with the sponsor; Liver transaminases (alanine aminotransferase [ALT])/aspartate aminotransferase [AST]) <=3.0*ULN.
5. Has recovered from adverse reactions to prior myeloma treatment or procedures (example, chemotherapy, immunotherapy, radiation therapy) to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0 Grade <=1 or baseline treatment or have the toxicity established as sequela, except for sensory or motor neuropathy, which should have recovered to Grade <=2 or baseline; ; (Grade 1 for the bortezomib arm).

Exclusion criteria:

1. Currently participating in another MM interventional study, including other clinical trials with investigational agents (including investigational vaccines or investigational medical device for disease under study) throughout the duration of this study.
2. Received previous treatment with modakafusp alfa.
3. Has a diagnosis of primary amyloidosis, Waldenström disease, monoclonal gammopathy of undetermined significance or smoldering MM per IMWG criteria or standard diagnostic criteria, plasma cell leukemia, POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes), lymphoplasmacytic lymphoma.
4. Has been diagnosed with another malignancy within the previous 3 years, except treated basal cell or localized squamous skin carcinomas, localized prostate cancer, cervical carcinoma in situ, resected colorectal adenomatous polyps, breast cancer in situ, or other malignancy for which the participant is not on active anticancer therapy and that in the opinion of the local investigator, with concurrence with the principal investigator, is considered cured with minimal risk of recurrence within 3 years.
5. Has evidence of central nervous system (CNS) involvement and/or meningeal involvement due to MM exhibited during screening.
6. Has a known severe allergic or anaphylactic reactions to human recombinant proteins or excipients used in the modakafusp alfa formulation or to the study combination agents, the study medications, their analogs, or excipients in the various formulations of any agent per the prescribing information.
7. Is seropositive for hepatitis B (defined by a positive test for hepatitis B surface antigen [HBsAg]). Participants with resolved infection (that is, participants who are HBsAg negative but positive for antibodies to hepatitis B core antigen and/or antibodies to hepatitis B surface antigen [anti-HBs]) must be screened using real-time polymerase chain reaction (PCR) measurement of hepatitis B virus (HBV) DNA levels. Those who are PCR positive will be excluded. EXCEPTION: Participants with serologic findings suggestive of HBV vaccination (anti-HBs positivity as the only serologic marker) and, a known history of prior HBV vaccination do not need to be tested for HBV DNA by PCR.
8. Has a known history of seropositivity for HIV.
9. Has a known history of seropositivity for hepatitis C (anti-hepatitis C virus [HCV] antibody positive or anti-hepatitis C virus-RNA quantitation positive). Exception: Participants with a sustained virologic response with undetectable HCV RNA level at least 12 weeks after completion of antiviral therapy.
10. For bortezomib arms: participants received a strong cytochromes P450 (CYP3A4) inducer within 5 half-lives prior to randomization.
11. The participant has a chronic condition requiring the use of systemic corticosteroids >10 mg/dL of prednisone or equivalent, in addition to any required corticosteroids for the treatment of MM.
12. Has a QTcF (QT interval corrected with Fridericia correction method >480 millisecond (ms) (Grade >=2).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2023-01-12 (Actual); Primary Completion 2024-06-04 (Actual); Study Completion 2024-06-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (21):
- United States (14):
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Scripps Health, San Diego, California
  - The University of Iowa Hospitals & Clinics, Iowa City, Iowa
  - Cancer Center At Greater Baltimore Medical Center, Baltimore, Maryland
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - NYU Langone Hospital - Long Island, Mineola, New York
  - New York University School of Medicine, New York, New York
  - Weill Cornell Medicine/New York Presbyterian Hospital, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Memorial Sloan Kettering Cancer Center - Main Campus, New York, New York
  - Novant Health Cancer Institute, Charlotte, North Carolina
  - Novant Health Cancer Institute - Forsyth Medical Center, Winston-Salem, North Carolina
  - Gabrail Cancer Center Research, Canton, Ohio
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
- Belgium (2):
  - CHU UCL Namur site Godinne, Yvoir, Namur
  - AZ Delta, Roeselare, Roeselare West-Vlaanderen
- Rambam Health Care Campus (RHCC) - Meyer Children's Hospital - Pediatric Diabetes & Obesity Clinic, Haifa, Israel
- Spain (4):
  - Clinica Universidad de Navarra-Sede Madrid, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Clinica Universidad de Navarra, Dept of Oncology, Pamplona
  - Hospital Universitario La Fe de Valencia, Valencia

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the study protocol and the statistical analysis plan. Requests will be assessed for scientific merit, product approval status, and conflicts of interest. If the request is approved, patient level data will be de-identified and study documents will be redacted to protect the privacy of trial participants and to protect commercially confidential information. Please visit USMedInfo@tevapharm.com to make your request.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at various investigative sites globally from 12 January 2023 to 04 June 2024.
Pre-assignment Details: Participants with a diagnosis of multiple myeloma (MM) were enrolled in this study. Participants with newly diagnosed MM (NDMM) received modakafusp alfa in combination with lenalidomide and participants with relapsed/refractory MM (RRMM) received modakafusp alfa in combination with pomalidomide or carfilzomib. Due to early termination of the study no participants were enrolled in Group 2 Arm 4: modakafusp alfa + bortezomib and Group 3 arms.
Groups:
- Group 3 (RRMM Triplets): Modakafusp Alfa + Pomalidomide + Bortezomib: Participants were planned to receive modakafusp alfa, infusion IV, once on Day 1, Q4W in combination with pomalidomide capsules orally once daily on Days 1 to 21 in a 28-day (4-week) treatment cycle along with bortezomib injection subcutaneously on Days 8, 15 and 22 for the first 8 cycles and subsequently on Days 8 and 22 of a 28-day (4-week) treatment cycle until disease progression, unacceptable toxicity, or until any other discontinuation criterion is met, whichever occurs first.
- Group 3 (RRMM Triplets): Modakafusp Alfa + Daratumumab + Pomalidomide: Participants were planned to receive modakafusp alfa, infusion IV, once on Day 1, Q4W in combination with daratumumab injection subcutaneously on Days 1, 8, 15 and 22 of Cycles 1 and 2, further followed by on Days 1 and 15 of Cycles 3 to 6, thereafter on Day 1 on a 28-day (4-week) treatment cycle along with pomalidomide capsules orally once daily on Days 1 to 21 in a 28-day (4-week) treatment cycle until disease progression, unacceptable toxicity, or until any other discontinuation criterion is met, whichever occurs first.
Period: Overall Study
Arm/Group | Group 1 (NDMM): Modakafusp Alfa 80 mg + Lenalidomide 10 mg | Group 2 (RRMM Doublets): Modakafusp Alfa 80 mg + Pomalidomide 2 mg | Group 2 (RRMM Doublets): Modakafusp Alfa 80 mg + Pomalidomide 4 mg | Group 2 (RRMM Doublets): Modakafusp Alfa 80 mg + Carfilzomib 20/70 mg/m^2 | Group 2 (RRMM Doublets) Arm 4: Modakafusp Alfa + Bortezomib | Group 3 (RRMM Triplets): Modakafusp Alfa + Pomalidomide + Bortezomib | Group 3 (RRMM Triplets): Modakafusp Alfa + Daratumumab + Pomalidomide
Started | 3 | 4 | 4 | 3 | 0 | 0 | 0
Completed | 2 | 1 | 2 | 2 | 0 | 0 | 0
Not Completed | 1 | 3 | 2 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 2 | 1 | 0 | 0 | 0
Not completed — Study Terminated by Sponsor | 0 | 3 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set (SAS) included all participants who had received at least 1 dose, even if incomplete, of any study drug. Due to early termination of the study no participants were enrolled in Group 2 Arm 4: modakafusp alfa + bortezomib and Group 3 arms, thus they are not presented here.
Groups:
- Group 1 (NDMM): Modakafusp Alfa 80 mg + Lenalidomide 10 mg: Participants received 80 mg modakafusp alfa, infusion IV, once on Day 1, Q4W, in combination with 10 mg lenalidomide capsules orally once daily continuously on Days 1 to 28, in a 28-day (4-week) treatment cycle until disease progression, unacceptable toxicity, or to a maximum of 2 years for MRD [-] negative participants, whichever occurred first.
- Group 2 (RRMM Doublets): Modakafusp Alfa 80 mg + Carfilzomib 20/70 mg/m^2: Participants received 80 mg modakafusp alfa, infusion IV, once on Day 1, Q4W in combination with 20/70 mg/m^2 carfilzomib IV, on Day 1, 8 and 15 of a 28-day (4-week) treatment cycle until disease progression, unacceptable toxicity, or until any other discontinuation criterion was met, whichever occurred first.
- Total: Total of all reporting groups
Arm/Group | Group 1 (NDMM): Modakafusp Alfa 80 mg + Lenalidomide 10 mg | Group 2 (RRMM Doublets): Modakafusp Alfa 80 mg + Pomalidomide 2 mg | Group 2 (RRMM Doublets): Modakafusp Alfa 80 mg + Pomalidomide 4 mg | Group 2 (RRMM Doublets): Modakafusp Alfa 80 mg + Carfilzomib 20/70 mg/m^2 | Total
Number analyzed (Participants) | 3 | 4 | 4 | 3 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.3 (18.50) | 64.3 (11.00) | 71.3 (2.63) | 57.3 (12.06) | 64.4 (11.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2 | 0 | 4
  Male | 1 | 4 | 2 | 3 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 2 | 4 | 3 | 11
  Unknown or Not Reported | 1 | 2 | 0 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 2 | 1 | 5
  White | 2 | 1 | 2 | 2 | 7
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose-limiting Toxicities (DLTs)
Description: DLT was defined by national cancer institute common terminology criteria for adverse events (NCI CTCAE) version 5.0: Grade 5 AE; Hematologic toxicity: Nonfebrile Grade 4 neutropenia lasting more than 7 consecutive days/Grade greater than or equal to (>=) 3 febrile neutropenia; Grade 4 thrombocytopenia lasting more than 14 consecutive days, Grade 3 thrombocytopenia with clinically significant bleeding; any other Grade 4 with exceptions; Nonhematologic Grade 3 or higher toxicities unrelated to the underlying disease with exceptions.
Time Frame: Cycle 1 (Cycle length is 28 days)
Population: The DLT-evaluable Analysis Set included participants who experienced a DLT in Cycle 1 in the treatment phase of the study or completed Cycle 1 procedures and received a full Cycle 1 dose of modakafusp alfa and at least 75% of the planned dose of the combination partner. Due to early termination of the study no participants were enrolled in Group 2 Arm 4: modakafusp alfa + bortezomib and Group 3 arms, thus they are not presented here.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (NDMM): Modakafusp Alfa 80 mg + Lenalidomide 10 mg | Group 2 (RRMM Doublets): Modakafusp Alfa 80 mg + Pomalidomide 2 mg | Group 2 (RRMM Doublets): Modakafusp Alfa 80 mg + Pomalidomide 4 mg | Group 2 (RRMM Doublets): Modakafusp Alfa 80 mg + Carfilzomib 20/70 mg/m^2
Number analyzed (Participants) | 2 | 3 | 4 | 2
Participants | 0 | 1 | 1 | 2

2. Primary Outcome: Number of Participants With One or More Treatment Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) is defined as any untoward medical occurrence in a participants administered a pharmaceutical product; the untoward medical occurrence does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product whether or not it is related to the medicinal product. A TEAE was any AE either reported for the first time or worsening of a pre-existing event after first dose of study drug and within 30 days of the last administration of study drug.
Time Frame: Up to 16.7 months
Population: The SAS included all participants who had received at least 1 dose, even if incomplete, of any study drug. Due to early termination of the study no participants were enrolled in Group 2 Arm 4: modakafusp alfa + bortezomib and Group 3 arms, thus they are not presented here.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (NDMM): Modakafusp Alfa 80 mg + Lenalidomide 10 mg | Group 2 (RRMM Doublets): Modakafusp Alfa 80 mg + Pomalidomide 2 mg | Group 2 (RRMM Doublets): Modakafusp Alfa 80 mg + Pomalidomide 4 mg | Group 2 (RRMM Doublets): Modakafusp Alfa 80 mg + Carfilzomib 20/70 mg/m^2
Number analyzed (Participants) | 3 | 4 | 4 | 3
Participants | 3 | 3 | 4 | 3

3. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as the time from the date on which the first dose of study drug is administered to the date of first documentation of confirmed progression of disease (PD) or death due to any cause, whichever occurs first. PD was determined by International Myeloma Working Group (IMWG) criteria. PD: increase of ≥25 percent (%) from lowest response value in any one or more of the following: serum M-component increase ≥0.5 gram per deciliter (g/dL) or urine M-component increase ≥200 milligram (mg)/24-hour; difference between involved and uninvolved free light chains (FLC) levels increase must be greater than (>) 10 milligram per deciliter (mg/dL); bone marrow plasma cell ≥10%; definite development of new bone lesions or soft tissue plasmacytomas or definite increase in the size of existing bone lesions or soft tissue plasmacytomas; development of hypercalcemia that can be attributed solely to plasma cell proliferative disorder.
Time Frame: Up to 16.7 months
Reporting Status: Not Posted

4. Secondary Outcome: Overall Response Rate (ORR)
Description: ORR: percentage of participants achieving confirmed partial response rate(PR)or better(stringent complete response[sCR]+complete response[CR]+very good partial response[VGPR]+PR)during study as defined by IMWG uniform response criteria and as determined by investigator.PR:>=50%reduction of serum M-protein and>=90% reduction in urine M-protein or less than(<)200mg/24 hour, or>=50%decrease in uninvolved FLC or >=50% reduction in plasma cells. At baseline,a >=50% decrease in size of soft tissue plasmacytomas was required. Percentages were rounded off to nearest single decimal place. Due to early termination of study no participants were enrolled in Group 2 Arm 4: modakafusp alfa+bortezomib and Group 3 arms, thus they are not presented here. Also, no participants in Group 1 fulfilled criteria for Response-Evaluable Analysis Set, hence are not presented here. Given limited number of participants and low confidence interval as a consequence, those response rate provides limited information.
Time Frame: Up to 16.7 months
Population: Response-Evaluable Analysis Set was a subset of SAS including participants with measurable disease at baseline & at least 1 post-baseline efficacy evaluation.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 2 (RRMM Doublets): Modakafusp Alfa 80 mg + Pomalidomide 2 mg | Group 2 (RRMM Doublets): Modakafusp Alfa 80 mg + Pomalidomide 4 mg | Group 2 (RRMM Doublets): Modakafusp Alfa 80 mg + Carfilzomib 20/70 mg/m^2
Number analyzed (Participants) | 4 | 4 | 3
percentage of participants | 0 [0.00 to 60.24] | 50 [6.76 to 93.24] | 33.3 [0.84 to 90.57]

5. Secondary Outcome: Duration of Response (DOR)
Description: DOR was defined as the time from the date of first documentation of confirmed PR or better (sCR+ CR+ VGPR+ PR) to the date of first documentation of PD or death due to any cause. PR: >=50% reduction of serum M-protein and >=90% reduction in urine M-protein or <200 mg/24 hour, or >=50% decrease in uninvolved FLC or >=50% reduction in plasma cells. At baseline, a >=50% decrease in size of soft tissue plasmacytomas is required. PD: increase of >=25% from lowest response value in any one or more of the following: serum M-component increase >=0.5 g/dL or urine M-component increase >=200 mg/24-hour; difference between involved and uninvolved FLC levels increase must be >10 mg/dL; bone marrow plasma cell >=10%; definite development of new bone lesions or soft tissue plasmacytomas or definite increase in the size of existing bone lesions or soft tissue plasmacytomas; development of hypercalcemia that can be attributed solely to plasma cell proliferative disorder.
Time Frame: Up to 16.7 months
Reporting Status: Not Posted

6. Secondary Outcome: Groups 2 and 3: Overall Survival (OS)
Description: OS was defined as the time from the first dose of administration to the date of death, due to any cause. Participants without documentation of death at the time of analysis were censored at the date last known to be alive.
Time Frame: Up to 16.7 months
Reporting Status: Not Posted

7. Secondary Outcome: Groups 2 and 3: Time to Progression (TTP)
Description: TTP was defined as the time from the date of the first dose until the earliest date of confirmed PD per IMWG, or death due to PD. PD: increase of >=25% from lowest response value in any one or more of the following: serum M-component increase >=0.5 g/dL or urine M-component increase >=200 mg/24-hour; difference between involved and uninvolved FLC levels increase must be >10 mg/dL; bone marrow plasma cell >=10%; definite development of new bone lesions or soft tissue plasmacytomas or definite increase in the size of existing bone lesions or soft tissue plasmacytomas; development of hypercalcemia that can be attributed solely to plasma cell proliferative disorder.
Time Frame: Up to 16.7 months
Reporting Status: Not Posted

8. Secondary Outcome: Groups 2 and 3: Time to Next Treatment (TTNT)
Description: TTNT was defined as the time from the date of first dose administration to the date of the first dose initiation of the next line of antineoplastic therapy, for any reason.
Time Frame: Up to 16.7 months
Reporting Status: Not Posted

9. Secondary Outcome: Groups 2 and 3: Disease Control Rate (DCR)
Description: DCR was defined as the percentage of participants who achieved a stable disease (SD) or better during the study based on the investigator's disease assessment as defined by IMWG uniform response criteria. SD was defined as no known evidence of progressive disease or new bone lesions. Percentages were rounded off to the nearest single decimal place.
Time Frame: Up to 16.7 months
Population: The Response-Evaluable Analysis Set was a subset of SAS including participants with measurable disease at baseline and at least 1 post-baseline efficacy evaluation. Due to early termination of the study no participants were enrolled in Group 2 Arm 4: modakafusp alfa + bortezomib and Group 3 arms, thus they are not presented here. Also, no participants in Group 1 fulfilled the criteria for the Response-Evaluable Analysis Set and hence are not presented here.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 2 (RRMM Doublets): Modakafusp Alfa 80 mg + Pomalidomide 2 mg | Group 2 (RRMM Doublets): Modakafusp Alfa 80 mg + Pomalidomide 4 mg | Group 2 (RRMM Doublets): Modakafusp Alfa 80 mg + Carfilzomib 20/70 mg/m^2
Number analyzed (Participants) | 4 | 4 | 3
percentage of participants | 75.0 [19.41 to 99.37] | 50.0 [6.76 to 93.24] | 66.7 [9.43 to 99.16]

10. Secondary Outcome: Groups 2 and 3: Event-free Survival (EFS)
Description: EFS was defined as the time from the date on which the first dose of study drug is administered to the date of the first documentation of an event that may include confirmed PD, discontinuation of a treatment for an AE (related or not related), or death due to any cause, whichever occurs first. PD was determined by IMWG criteria. PD: increase of >=25 % from lowest response value in any one or more of the following: serum M-component increase >=0.5 g/dL or urine M-component increase >=200 mg/24-hour; difference between involved and uninvolved FLC levels increase must be > 10 mg/dL; bone marrow plasma cell >=10%; definite development of new bone lesions or soft tissue plasmacytomas or definite increase in the size of existing bone lesions or soft tissue plasmacytomas; development of hypercalcemia that can be attributed solely to plasma cell proliferative disorder.
Time Frame: Up to 16.7 months
Reporting Status: Not Posted

11. Secondary Outcome: Groups 2 and 3: Time to Response (TTR)
Description: TTR was defined as the time from the date of the first dose administration to the date of the first documentation of objective confirmed response as defined by IMWG criteria.
Time Frame: Up to 16.7 months
Reporting Status: Not Posted

12. Secondary Outcome: Group 1: Percentage of Participants With MRD Negativity Status at a Threshold of 10^-5
Description: Rate of MRD negativity at a sensitivity of 10^-5 was defined as the percentage of participants who achieved MRD negative status in the MRD-evaluable analysis set.
Time Frame: At 6 months, 1 year, and 2 years after the start of treatment
Population: MRD data was not collected as no participant achieved the criteria for MRD-evaluable analysis set (i.e., being on study at 6 months).
Arm/Group | Group 1 (NDMM): Modakafusp Alfa 80 mg + Lenalidomide 10 mg
Number analyzed (Participants) | 0

13. Secondary Outcome: Groups 2 and 3: Percentage of Participants With MRD Negativity CR Status at a Threshold of 10^-5 in Participants Achieving CR Assessed by the Investigator
Description: Rate of MRD negativity CR status a sensitivity of 10^-5 was defined as the percentage of participants who have achieved MRD negative CR status in participants achieving CR. CR is defined as negative immunofixation of serum and urine, disappearance of any soft tissue plasmacytomas, and <5% plasma cells in bone marrow; in participants for whom only measurable disease is by serum FLC level, normal FLC ratio of 0.26 to 1.65 in addition to CR criteria is required.
Time Frame: Up to 2 years after CR confirmation
Population: MRD data was not collected as no participant achieved the criteria for MRD-evaluable analysis set (i.e., achieving a Complete Response).
Arm/Group | Group 2 (RRMM Doublets): Modakafusp Alfa 80 mg + Pomalidomide 2 mg | Group 2 (RRMM Doublets): Modakafusp Alfa 80 mg + Pomalidomide 4 mg | Group 2 (RRMM Doublets): Modakafusp Alfa 80 mg + Carfilzomib 20/70 mg/m^2
Number analyzed (Participants) | 0 | 0 | 0

14. Secondary Outcome: Duration of MRD Negativity Status at a Threshold of 10^-5 in Participants Achieving MRD Negativity
Description: Duration of MRD negativity (10^-5) was defined as the time from the date of first documentation of MRD[-] to the first documentation of MRD positivity or confirmed PD or death due to any cause, whichever occurred first. PD: increase of >=25% from lowest response value in any one or more of the following: serum M-component increase >=0.5 g/dL or urine M-component increase >=200 mg/24-hour; difference between involved and uninvolved FLC levels increase must be >10 mg/dL; bone marrow plasma cell >=10%; definite development of new bone lesions or soft tissue plasmacytomas or definite increase in the size of existing bone lesions or soft tissue plasmacytomas; development of hypercalcemia that can be attributed solely to plasma cell proliferative disorder.
Time Frame: Up to 2 years after treatment
Population: as for outcome 13
Arm/Group | Group 1 (NDMM): Modakafusp Alfa 80 mg + Lenalidomide 10 mg | Group 2 (RRMM Doublets): Modakafusp Alfa 80 mg + Pomalidomide 2 mg | Group 2 (RRMM Doublets): Modakafusp Alfa 80 mg + Pomalidomide 4 mg | Group 2 (RRMM Doublets): Modakafusp Alfa 80 mg + Carfilzomib 20/70 mg/m^2
Number analyzed (Participants) | 0 | 0 | 0 | 0

15. Secondary Outcome: Group 2 and 3: Percentage of Participants With MRD Negativity Status at a Threshold of 10^-5
Description: Rate of MRD negativity at a sensitivity of 10^-5 was defined as the percentage of participants who have achieved MRD negative status.
Time Frame: Up to 16.7 months
Population: as for outcome 13
Arm/Group | Group 2 (RRMM Doublets): Modakafusp Alfa 80 mg + Pomalidomide 2 mg | Group 2 (RRMM Doublets): Modakafusp Alfa 80 mg + Pomalidomide 4 mg | Group 2 (RRMM Doublets): Modakafusp Alfa 80 mg + Carfilzomib 20/70 mg/m^2
Number analyzed (Participants) | 0 | 0 | 0

16. Secondary Outcome: Groups 2 and 3: Duration of MRD Negativity Status at a Sensitivity Threshold of 10^-5 in Participants Achieving MRD Negativity
Description: as for outcome 14
Time Frame: Up to 16.7 months
Population: as for outcome 13
Arm/Group | Group 2 (RRMM Doublets): Modakafusp Alfa 80 mg + Pomalidomide 2 mg | Group 2 (RRMM Doublets): Modakafusp Alfa 80 mg + Pomalidomide 4 mg | Group 2 (RRMM Doublets): Modakafusp Alfa 80 mg + Carfilzomib 20/70 mg/m^2
Number analyzed (Participants) | 0 | 0 | 0

17. Secondary Outcome: Number of Participants With Positive Anti-drug Antibodies (ADA) and Neutralizing Antibody (NAb)
Time Frame: Up to 16.7 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 16.7 months
Description: The SAS included all participants who had received at least 1 dose, even if incomplete, of any study drug.
Arm/Group | Group 1 (NDMM): Modakafusp Alfa 80 mg + Lenalidomide 10 mg | Group 2 (RRMM Doublets): Modakafusp Alfa 80 mg + Pomalidomide 2 mg | Group 2 (RRMM Doublets): Modakafusp Alfa 80 mg + Pomalidomide 4 mg | Group 2 (RRMM Doublets): Modakafusp Alfa 80 mg + Carfilzomib 20/70 mg/m^2
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/4 | 2/4 | 1/3
Serious Adverse Events (participants affected / at risk) | 0/3 | 1/4 | 1/4 | 3/3
Other Adverse Events (participants affected / at risk) | 3/3 | 3/4 | 4/4 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 (NDMM): Modakafusp Alfa 80 mg + Lenalidomide 10 mg (N=3) | Group 2 (RRMM Doublets): Modakafusp Alfa 80 mg + Pomalidomide 2 mg (N=4) | Group 2 (RRMM Doublets): Modakafusp Alfa 80 mg + Pomalidomide 4 mg (N=4) | Group 2 (RRMM Doublets): Modakafusp Alfa 80 mg + Carfilzomib 20/70 mg/m^2 (N=3)
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Haemolytic uraemic syndrome (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 1
Pneumonia influenzal (Infections and infestations) | 0 | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 1
Renal haemorrhage (Renal and urinary disorders) | 0 | 0 | 0 | 1
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 (NDMM): Modakafusp Alfa 80 mg + Lenalidomide 10 mg (N=3) | Group 2 (RRMM Doublets): Modakafusp Alfa 80 mg + Pomalidomide 2 mg (N=4) | Group 2 (RRMM Doublets): Modakafusp Alfa 80 mg + Pomalidomide 4 mg (N=4) | Group 2 (RRMM Doublets): Modakafusp Alfa 80 mg + Carfilzomib 20/70 mg/m^2 (N=3)
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 2
Anaemia (Blood and lymphatic system disorders) | 2 | 2 | 3 | 3
Anal incontinence (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 2
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 1
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 2 | 0
Bradycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Bundle branch block left (Cardiac disorders) | 0 | 0 | 0 | 1
Chills (General disorders) | 0 | 0 | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Ear infection (Infections and infestations) | 0 | 1 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 1
Fatigue (General disorders) | 1 | 2 | 2 | 0
Gastroenteritis salmonella (Infections and infestations) | 0 | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Haematoma (Vascular disorders) | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypogammaglobulinaemia (Immune system disorders) | 0 | 0 | 2 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2
Inflammation (General disorders) | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 2
Leukopenia (Blood and lymphatic system disorders) | 2 | 0 | 0 | 0
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 1 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 3 | 3 | 3 | 0
Noninfective sialoadenitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 1
Portal hypertension (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 1 | 0 | 1
Rhinitis (Infections and infestations) | 0 | 1 | 0 | 0
Right ventricular dysfunction (Cardiac disorders) | 0 | 0 | 0 | 1
Sacral pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Salmonella bacteraemia (Infections and infestations) | 0 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 1
Suprapubic pain (General disorders) | 0 | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 3 | 3 | 3
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
Study was terminated early by sponsor for strategic reasons. No participants were enrolled in Group 2 Arm 4: modakafusp alfa + bortezomib & Group 3 arms. Data for endpoints related to PFS, OS, DOR, TTP, TTNT, EFS, TTR, & MRD were not collected as planned & hence not reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2024-09-19): https://cdn.clinicaltrials.gov/large-docs/16/NCT05556616/Prot_000.pdf
  • Statistical Analysis Plan (2022-05-09): https://cdn.clinicaltrials.gov/large-docs/16/NCT05556616/SAP_001.pdf